CLINICAL TRIAL: NCT02613247
Title: Intra-articular Hyaluronic Acid Injection for Therapy-resistant Patellofemoral Pain Syndrome: an Open-label, Randomized, Delayed-start Clinical Trial
Brief Title: Intra-articular Hyaluronic Acid Injection for Therapy-resistant Patellofemoral Pain Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Jordan Raugust, Principal Investigator, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VIP-123
Record Dates: First submitted 2015-11-20; First posted 2015-11-24 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: Viscosupplementation; Hyaluronic acid; Synvisc; Synvisc-One; Patellofemoral pain syndrome; PFPS; Anterior knee pain; Runner's knee
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate-start group (Experimental): Hylan G-F 20 6 mL intra-articular knee injection
  Interventions: Device: Hylan G-F 20
- Delayed-start group (Other): Washout control group which then becomes an experimental group (Hylan G-F 20 6 mL intra-articular knee injection) at 6 weeks post-enrolment
  Interventions: Device: Hylan G-F 20

INTERVENTIONS:
Device: Hylan G-F 20 — Intra-articular injection of 6 mL Hylan G-F 20
  Other Names: Synvisc-One

SUMMARY:
Patellofemoral pain syndrome (PFPS) is the most common overuse injury seen in the athletic population, particularly amongst runners. The standard of care treatment for PFPS is a comprehensive active rehabilitation program. Eighty percent of patients with PFPS report improvement in their symptoms with such a program. Unfortunately, the remaining twenty percent fail to achieve adequate symptom relief with rehabilitation alone. Considering the enormous number of individuals running for fitness, PFPS represents a significant challenge to public health as the investigators strive to encourage active living in our society.

A relationship between PFPS and the development of patellofemoral osteoarthritis (PFOA) has been suggested in scientific literature. Given that intra-articular viscosupplementation (hyaluronic acid) injections have shown clinically significant symptom improvement in knee osteoarthritis, and PFPS is likely on the same spectrum, the investigators propose a trial for therapy-resistant PFPS.

Hyaluronic acid is a naturally occurring molecule found in the synovial fluid of freely movable joints (such as the knee). It is believed to contribute to lubrication and cushioning in these joints. The composition of synovial fluid within arthritic joints is altered, resulting in reduced fluid viscosity and elasticity. One modern formulation of hyaluronic acid is Hylan G-F 20 (Synvisc-One, Sanofi Canada). This treatment is offered as a single injection and will be utilized in this clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18-45
2. Previously diagnosed with PFPS that failed to improve with at least 6 weeks of active rehabilitation, supervised by physiotherapist.
3. Retropatellar or peripatellar knee pain for a minimum of 2 months
4. Pain aggravated by at least two of the following patellofemoral joint loading activities: squatting, running, ascending or descending stairs, or sitting with prolonged knee flexion
5. Pain with patellar grind test on clinical examination
6. Visual Analog Scale (VAS) > 4/10 with patellofemoral joint loading activities
7. Normal knee x-ray

Exclusion Criteria:

1. X-ray evidence of osteoarthritis or fracture
2. Meniscal or ligamentous injury suspected clinical examination
3. Previous knee surgery
4. History of patellar instability or positive patellar apprehension test
5. Any contraindication to knee injection (overlying skin or joint infection, joint effusion, coagulopathy, previous adverse reaction etc.)
6. Known allergy to avian products
7. Previous knee injection within the last 3 months
8. Pregnant or breastfeeding

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Pain measured using the visual analog scale (VAS) | 6 weeks

SECONDARY OUTCOMES:
Function measured using the Anterior Knee Pain Scale (AKPS) | 6 weeks and 12 weeks
Pain measured using the visual analog scale (VAS) | Weekly until 12 weeks post injection
Kinetic and kinematic data | Baseline compared to 6 weeks post injection
  Data will be collected using a 3-D motion analysis system with 8 cameras and an instrumented treadmill

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Raugust, Principal Investigator — University of Calgary; Andrew Malawski, Study Director — University of Calgary; Reed Ferber, Study Chair — University of Calgary
Locations (1):
- Calgary Running Injury Clinic, Calgary, Alberta, Canada